CLINICAL TRIAL: NCT01201174
Title: Oxidative Stress Contributes to Hemolysis in Patients With Hereditary Spherocytosis (HS) and Can be Ameliorated by Fermented Papaya Preparation (FPP)
Brief Title: Hemolysis in Patients With Hereditary Spherocytosis (HS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dr. Ghoti Hossam, Organization: hematology department on Wolfsson Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SH-01CTIL
Record Dates: First submitted 2010-09-12; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Hereditary; Hemolysis
Keywords: Hemolysis in Patients with Hereditary Spherocytosis; with documented family history of HS.; spherocyte morphology,; splenomegaly and non-immune mediated hemolysis.
MeSH Terms: conditions — Hemolysis; Splenomegaly | interventions — fermented papaya preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with Hereditary Spherocytosis (No Intervention): All patients should have clinical and laboratory findings, consistent with mild to severe HS, diagnosed on the basis of spherocyte morphology, elevated MCHC (33-38 g/dl), with a mean value of (35.47 g/dl), increased osmotic fragility , splenomegaly and non-immune mediated hemolysis.
  Interventions: Other: fermented papaya preparation (FPP)

INTERVENTIONS:
Other: fermented papaya preparation (FPP) — Hemolysis will be assayed by suspending 3 ml of packed RBC in PBS or in the autologous plasma and overnight incubation in the presence of various concentrations of antioxidants such as fermented papaya preparation (FPP) at 37oC in humidified atmosphere of 5% CO2 in air (10). Following 5 min centrifugation at 800 rpm, the supernatants will collected for Hb determination by measuring the absorbance at 540 nm.

SUMMARY:
In the present study the investigators are going to explore the oxidative status of HS-RBC and its contribution to hemolysis

DETAILED DESCRIPTION:
The oxidative status of cells, which is determined by the balance between pro-oxidants, such as the reactive oxygen species (ROS), and antioxidants, is a major regulator of cellular functions. Impaired balance between pro- and antioxidants causes oxidative stress which may result in oxidation of proteins, lipids and DNA with the final outcome of premature cell aging and apoptosis [1,2]. Oxidatively stressed red blood cell (RBC) have been observed in various congenital and acquired hemolytic anemias, including thalassemia, sickle cell anemia, congenital dyserythropoietic anemia, G6PD deficiency and paroxysmal nocturnal hemoglobinuria (PNH) as well as in myelodysplastic syndrome (MDS). Although the primary etiology is different in these anemias, oxidative stress mediates several of their pathologies, mainly hemolysis [3].

Hereditary Spherocytosis (HS) is a genetic disorder of the RBC skeleton with primary deficiency in spectrin, ankyrin-1, band 3 or protein 4.2 associated with chronic hemolytic anemia [4]. Secondary protein deficiencies resulting from oxidative stress are often observed and may be involved in the clinical manifestations of the disease [5].

ELIGIBILITY:
Inclusion Criteria:

* patients > 5 years
* with documented family history of HS
* patients should have clinical and laboratory findings, consistent with mild to severe HS, diagnosed on the basis of spherocyte morphology, elevated MCHC (33-38 g/dl), with a mean value of (35.47 g/dl), increased osmotic fragility , splenomegaly and non-immune mediated hemolysis.

Exclusion Criteria:

* non

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
ROS, reduced glutathione (GSH) and lipid peroxides will be measured in RBC | year
  ROS, reduced glutathione (GSH) and lipid peroxides will be measured in RBC following incubation with with 100 μM 2'-7'-dichlorofluorescin diacetate, 40 μM [1-(4-chloromercuryphenyl-azo-2-naphthol)] and fluor-DHPE, respectively for ROS [8] and with mercury orange for GSH [9]. After being washed twice, the cells will be resuspended in PBS and analyzed by flow cytometry .

SECONDARY OUTCOMES:
Hemolysis | year
  Hemolysis will be assayed by suspending 3 ml of packed RBC in PBS or in the autologous plasma and overnight incubation in the presence of various concentrations of antioxidants such as fermented papaya preparation (FPP)

CONTACTS AND LOCATIONS:
Overall Officials: GHOTI HOSSAM, doctor, Principal Investigator — HEMATOLOGY DEPARTMENT ON WOLFSSON MEDICAL CENTER
Locations (1):
- Wolfsson Medical Center, Holon, Israel,, Israel